CLINICAL TRIAL: NCT01507896
Title: BAX 326 (Recombinant Factor IX): A Phase 3 Prospective, Multicenter Study Evaluating Efficacy and Safety in Previously Treated Patients With Severe (FIX Level < 1%) or Moderately Severe (FIX Level 1-2%) Hemophilia B Undergoing Surgical or Other Invasive Procedures
Brief Title: BAX 326 Surgery Study in Hemophilia B Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 251002; 2011-000413-39 (EudraCT Number)
Record Dates: First submitted 2012-01-09; First posted 2012-01-11 (Estimated); Results first posted 2017-02-15 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Hemophilia B
MeSH Terms: conditions — Hemophilia B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BAX326 in Surgery (Experimental): BAX 326 (recombinant factor IX) in Surgery
  Interventions: Biological: Recombinant factor IX

INTERVENTIONS:
Biological: Recombinant factor IX — Following a loading dose with BAX326, participants will receive BAX326 as a bolus infusion. The treatment regimen will be determined by the intensity and duration of the hemostatic challenge and the institution´s standard of care. The dose will be tailored to raise FIX concentration to at least 80%-100% of normal for major surgeries and to at least 30%-60% of normal for minor surgeries.
  Other Names: BAX326; RIXUBIS

SUMMARY:
The purpose of the study is to assess the hemostatic efficacy and safety of BAX 326 in subjects with severe (FIX level < 1%) or moderately severe (FIX level 1-2%) hemophilia B undergoing major or minor elective or emergency surgical, dental or other invasive procedures.

ELIGIBILITY:
Main Inclusion Criteria:

* Participant and/or legal representative has/have voluntarily provided signed informed consent.
* Participant has severe (FIX level < 1%) or moderately severe (FIX level 1-2%) hemophilia B (based on the one stage activated partial thromboplastin time (aPTT) assay), as tested at screening at the central laboratory.
* Participant requires surgery
* Participant has previously been treated with plasma-derived and/or recombinant FIX concentrate(s) for a minimum of 150 exposure days
* Participant has no evidence of a history of FIX inhibitors
* Participant is immunocompetent as evidenced by a CD4 count ≥ 200 cells/mm3.
* Participant is human immunodeficiency (HIV) negative or is HIV+ with a viral load < 200 particles/μL ~ < 400,000 copies/mL.

Main Exclusion Criteria:

* Participant has a history of FIX inhibitors with a titer ≥ 0.6 Bethesda Units (BU) (as determined by the Nijmegen modification of the Bethesda assay or the assay employed in the respective local laboratory) at any time prior to screening.
* Participant has a detectable FIX inhibitor at screening, with a titer ≥0.6 Bethesda Units (BU) as determined by the Nijmegen modification of the Bethesda assay in the central laboratory.
* Participant has a history of allergic reaction or evidence of an ongoing or recent thrombotic disease, fibrinolysis or disseminated intravascular coagulation (DIC).
* Known hypersensitivity to hamster proteins or recombinant furin.
* Evidence of an ongoing or recent thrombotic disease, fibrinolysis or disseminated intravascular coagulation (DIC).
* Abnormal renal function
* Severe chronic liver disease
* Active hepatic disease with ALT or AST levels > 5 times the upper limit of normal.
* Diagnosis of an iherited or acquired hemostatic defect other than hemophilia B.
* Platelet count < 100,000/mL.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-12-19 (Actual); Primary Completion 2014-05-15 (Actual); Study Completion 2014-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (14):
- Instituto de Hematología y Medicina Clínica Rubén Dávoli, Rosario, Argentina
- Specialized Haematological Hospital "Joan Pavel", Sofia, Bulgaria
- Hospital Dr. Sotero del Rio, Santiago, Chile
- Centro Medico Imbanaco, Cali, Colombia
- Klinika detska hematologie a onkologie, Fakultni Nemocnice Motol, Prague, Czechia
- Poland (3):
  - Medical University Lodz, Copernicus Hospital, Department of Hematology, Lodz
  - Independent Public Pediatric Teaching Hospital, Clinical Department of Hematology and Pediatrics, Warsaw
  - Institute of Haematology and Transfusion Medicine, Warsaw
- Louis Turcanu Emergency Clinical Children´s Hospital, Timișoara, Romania
- Russia (3):
  - Federal State Institution Kirov, Hematology and Blood Transfusion Research Institute under the Federal Agency for High-Tech Medical Care, Kirov
  - Children's Territorial Clinical Hospital, Krasnodar
  - Hematology Research Center RAMS, Moscow
- State Institution "Institute of Blood Pathology and Transfusion Medicine under the Academy of Medical Sciences of Ukraine", Lviv, Ukraine
- Royal Manchester Children's Hospital, Department of Hematology, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Result] Windyga J, Lissitchkov T, Stasyshyn O, Mamonov V, Ghandehari H, Chapman M, Fritsch S, Wong WY, Pavlova BG, Abbuehl BE. Efficacy and safety of a recombinant factor IX (Bax326) in previously treated patients with severe or moderately severe haemophilia B undergoing surgical or other invasive procedures: a prospective, open-label, uncontrolled, multicentre, phase III study. Haemophilia. 2014 Sep;20(5):651-8. doi: 10.1111/hae.12419. Epub 2014 Apr 3. PMID 24697870
- [Derived] Windyga J, Timofeeva M, Stasyshyn O, Mamonov V, Lamas Castellanos JL, Lissitchkov T, Chojnowski K, Chapman M, Pavlova BG, Tangada S. Phase 3 Clinical Trial: Perioperative Use of Nonacog Gamma, a Recombinant Factor IX, in Previously Treated Patients With Moderate/Severe Hemophilia B. Clin Appl Thromb Hemost. 2020 Jan-Dec;26:1076029620946839. doi: 10.1177/1076029620946839. PMID 32816519

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was conducted at 10 clinical sites in 8 countries (Bulgaria, Czech Republic, Poland, Romania, Russia, Ukraine, Chile, Colombia).
Pre-assignment Details: 30 unique participants enrolled for 41 surgical procedures, of which 1 participant discontinued before treatment with BAX326 but re-enrolled later for another surgical procedure. Note: a unique participant can undergo more than one surgical procedure.
Groups:
- Treatment With BAX326: Recombinant Factor IX (FIX): Following a loading dose with BAX326, participants received BAX326 as a bolus infusion. The treatment regimen was determined by the intensity and duration of the hemostatic challenge and the institution's standard of care. The dose was tailored to raise FIX concentration to at least 80%-100% of normal for major surgeries and to at least 30%-60% of normal for minor surgeries. Note: Treatment with BAX326 refers to unique participants treated with BAX326 which is less than the number of participants treated with BAX326 as unique participants could undergo more than one surgical procedure in this study. 30 unique participants were treated with BAX326 for 40 planned surgical procedures; of these, 2 unique participants were treated with BAX326 but did not undergo 2 surgical procedures (1 surgery per unique participant), therefore 28 unique participants underwent 38 surgical procedures.
Period: Overall Study
Arm/Group | Treatment With BAX326
Started | 30 (30 unique participants had 40 surgeries planned (participants could have multiple surgeries).)
Completed | 28 (28 unique participants had 38 surgeries (participants could have multiple surgeries).)
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — The surgery was denied by the sponsor. | 1

BASELINE CHARACTERISTICS:
Population: Note there were 30 unique participants with a total of 40 planned surgeries, as participants may have > 1 surgery. Baseline data reflects number of planned surgeries.
Arm/Group | Treatment With BAX326
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.7 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 40

OUTCOME MEASURES:

1. Primary Outcome: Intraoperative Hemostatic Efficacy
Description: Assessment by the operating surgeon on a 4 point ordinal scale (according to the definitions provided below): - Excellent: Intraoperative blood loss was less than or equal to that expected for the type of procedure performed in a hemostatically normal participant (≤ 100% ) - Good: Intraoperative blood loss was up to 50% more than expected for the type of procedure performed in a hemostatically normal participant (101 - 150%) - Fair: Intraoperative blood loss was more than 50% of that expected for the type of procedure performed in a hemostatically normal participant (> 150%) - None: Uncontrolled hemorrhage that was the result of inadequate therapeutic response despite proper dosing, necessitating a change of Factor IX concentrate
Time Frame: On day of surgery
Population: All participants in the Full Analysis Set (participants exposed to BAX326 and provided data suitable for hemostatic efficacy analysis) treated with BAX326 and had surgery. Note: a unique participant could have more than one surgical procedure.
Measure: Number; unit: surgeries
Units Other Than Participants: surgeries
Groups:
- All Surgeries: All participants treated with BAX326 per surgical procedure. Data is reported per number of surgical procedures as opposed to number of unique participants as a unique participant can have more than one surgical procedure.
- Major Surgeries: Major surgery defined as surgeries which required moderate or deep sedation, general anesthesia, or major conduction blockade for patient comfort. It generally referred to major orthopedic (e.g., joint replacement), major abdominal, intracranial, cardiovascular, spinal and any other surgery which had a significant risk of large volume blood loss or blood loss into a confined anatomical space. Several tooth extractions or extraction of the third molar were generally considered as major.
- Minor Surgeries: Minor surgery defined as surgeries which could be safely and comfortably performed on a patient who had received local or topical anesthesia, without more than minimal pre-operative medication or minimal pre-operative medication or minimal intraoperative sedation. The likelihood of complications requiring hospitalization or prolonged hospitalization was remote. It referred to interventions such as removal of skin lesions, arthroscopy, minor dental procedures or dental extractions.
Arm/Group | All Surgeries | Major Surgeries | Minor Surgeries
Number analyzed (Participants) | 28 | 17 | 13
Number analyzed (surgeries) | 38 | 21 | 17
surgeries
  Excellent | 37 | 20 | 17
  Good | 1 | 1 | 0
  Fair | 0 | 0 | 0
  None | 0 | 0 | 0

2. Primary Outcome: Actual Intraoperative Blood Loss
Description: Actual intraoperative blood loss was determined by the drainage volume, if a drain was placed, and the estimated blood loss into swabs and towels during the procedure.
Time Frame: On day of surgery
Population: All participants in the Full Analysis Set (participants exposed to BAX326 and provided data suitable for hemostatic efficacy analysis) treated with BAX326 per surgical procedure. Note: a unique participant could have more than one surgical procedure.
Measure: Mean (Standard Deviation); unit: mL
Units Other Than Participants: surgeries
Arm/Group | All Surgeries | Major Surgeries | Minor Surgeries
Number analyzed (Participants) | 28 | 17 | 13
Number analyzed (surgeries) | 38 | 21 | 17
mL | 191.1 (354.1) | 344.9 (420.1) | 1.2 (1.1)

3. Primary Outcome: Actual Intraoperative Blood Loss Compared to Average and Maximum Blood Loss Predicted Preoperatively by the Operating Surgeon
Description: Predicted average/maximum blood loss minus actual blood loss. Prior to the surgery, the surgeon predicted the estimated volume (mL) of the expected average and maximum blood loss for the planned surgical intervention in a hemostatically normal individual of the same sex, age, and stature as the study participant for the intraoperative period.
Time Frame: On day of surgery
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL
Units Other Than Participants: surgeries
Arm/Group | All Surgeries | Major Surgeries | Minor Surgeries
Number analyzed (Participants) | 28 | 17 | 13
Number analyzed (surgeries) | 38 | 21 | 17
mL
  Difference from predicted average blood loss | -27.0 (158.9) | -50.9 (213.0) | 2.4 (4.9)
  Difference from predicted maximum blood loss | 128.3 (260.8) | 222.0 (323.7) | 12.5 (24.5)

4. Primary Outcome: Postoperative Hemostatic Efficacy at Drain Removal
Description: The postoperative hemostatic efficacy was to be assessed by the operating surgeon according to the following criteria (4-point ordinal scale): - Excellent: Volume in drain was less than or equal than that expected for the type of procedure performed in a hemostatically normal participant (≤ 100% ) - Good: Volume in drain was up to 50% more than expected for the type of procedure performed in a hemostatically normal participant (101% - 150%) - Fair: Volume in drain was more than 50% of that expected for the type of procedure performed in a hemostatically normal participant (> 150%) - None: Uncontrolled bleeding that was the result of inadequate therapeutic response despite proper dosing, necessitating a change of Factor IX concentrate
Time Frame: At drain removal (from 1-3 days postoperatively)
Population: Participants in the Full Analysis Set (participants exposed to BAX326 and provided data suitable for hemostatic efficacy analysis) who had a drain placed during surgery (major surgeries only). Note: a unique participant could have more than one surgical procedure
Measure: Number; unit: major surgeries with drain placed
Units Other Than Participants: major surgeries with drain placed
Groups:
- Major Surgeries: Major surgery defined as surgeries which required moderate or deep sedation, general anesthesia, or major conduction blockade for patient com fort. It generally referred to major orthopedic (e.g., joint replacement), major abdom inal, intracranial, cardiovascular, spinal and any other surgery which had a significant risk of large volume blood loss or blood loss into a confined anatom ical space. Several tooth extractions or extraction of the third molar were generally considered as major.
Arm/Group | Major Surgeries
Number analyzed (Participants) | 11
Number analyzed (major surgeries with drain placed) | 14
major surgeries with drain placed
  Excellent | 10
  Good | 4
  Fair | 0
  None | 0

5. Primary Outcome: Postoperative Hemostatic Efficacy at Postoperative Day 3
Description: Assessment by the operating surgeon on a 4 point ordinal scale: - Excellent: Postoperative hemostasis achieved with BAX326 was as good or better than that expected for the type of surgical procedure performed in a hemostatically normal participant - Good: Postoperative hemostasis achieved with BAX326 was probably as good as that expected for the type of surgical procedure performed in a hemostatically normal participant - Fair: Postoperative hemostasis with BAX326 was clearly less than optimal for the type of procedure performed but was maintained without the need to change the Factor IX concentrate - None: Participant experienced uncontrolled bleeding that was the result of inadequate therapeutic response despite proper dosing, necessitating a change of Factor IX concentrate
Time Frame: At postoperative day 3 (approximately 72 hours postoperatively)
Population: Participants in the Full Analysis Set who were provided with a hemostatic efficacy assessment by the operating surgeon at post operative day 3 where no drain was employed. Note: a unique participant could have more than one surgical procedure.
Measure: Number; unit: surgeries
Units Other Than Participants: surgeries
Arm/Group | All Surgeries | Major Surgeries | Minor Surgeries
Number analyzed (Participants) | 6 | 6 | 1
Number analyzed (surgeries) | 8 | 7 | 1
surgeries
  Excellent | 7 | 6 | 1
  Good | 1 | 1 | 0
  Fair | 0 | 0 | 0
  None | 0 | 0 | 0

6. Primary Outcome: Postoperative Hemostatic Efficacy on Day of Discharge
Description: as for outcome 5
Time Frame: At discharge from hospital (from 1-3 days postoperatively for minor surgery and approximately 2 weeks postoperatively for major surgery)
Population: as for outcome 2
Measure: Number; unit: surgeries
Units Other Than Participants: surgeries
Groups:
- All Surgical Procedures: All participants treated with BAX326 per surgical procedure. Data is reported per number of surgical procedures as opposed to number of unique participants as a unique participant can have more than one surgical procedure.
Arm/Group | All Surgical Procedures | Major Surgeries | Minor Surgeries
Number analyzed (Participants) | 28 | 17 | 13
Number analyzed (surgeries) | 38 | 21 | 17
surgeries
  Excellent | 29 | 12 | 17
  Good | 7 | 7 | 0
  Fair | 2 | 2 | 0
  None | 0 | 0 | 0

7. Primary Outcome: Actual Postoperative Blood Loss
Description: Postoperative blood loss was based on the drainage fluid and was only assessed for participants who had a drain placed during surgery.
Time Frame: At drain removal (from 1-3 days postoperatively)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mL
Units Other Than Participants: surgeries with drain placed
Arm/Group | Major Surgeries
Number analyzed (Participants) | 11
Number analyzed (surgeries with drain placed) | 14
mL | 603.6 (388.7)

8. Primary Outcome: Actual Postoperative Blood Loss Compared to Average and Maximum Blood Loss Predicated Preoperatively by the Operating Surgeon
Description: Predicted average/maximum blood loss minus actual blood loss for participants who had a drain placed during surgery. Prior to the surgery, the surgeon will predict the estimated volume (mL) of the expected average and maximum blood loss for the planned surgical intervention in a hemostatically normal individual of the same sex, age, and stature as the study subject for the postoperative period until drain removal.
Time Frame: At postoperative day 3 (approximately 72 hours postoperatively)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mL
Units Other Than Participants: surgeries with drain placed
Arm/Group | Major Surgeries
Number analyzed (Participants) | 11
Number analyzed (surgeries with drain placed) | 14
mL
  Difference from predicated average blood loss | -221.4 (331.7)
  Difference from predicted maximum blood loss | 147.1 (330.1)

9. Primary Outcome: Daily Weight-Adjusted Dose of BAX326 Per Participant
Description: Daily weight-adjusted doses of BAX326 per participant were recorded from the day of surgery until postoperative Days 11+. Each category in outcome measure includes number of all, major and minor surgeries, respectively, if different from the totals.
Time Frame: From initiation of surgery until discharge from hospital (from 1-3 days postoperatively for minor surgery and approximately 2 weeks postoperatively for major surgery)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: IU/kg
Units Other Than Participants: surgeries
Arm/Group | All Surgeries | Major Surgeries | Minor Surgeries
Number analyzed (Participants) | 28 | 17 | 13
Number analyzed (surgeries) | 38 | 21 | 17
IU/kg
  Day of Surgery | 144.8 (70.3) | 191.5 (50.6) | 87.2 (42.9)
  Postoperative Day 1 | 103.9 (44.6) | 136.7 (30.1) | 63.5 (18.0)
  Postoperative Day 2 (N=29,21,8) | 115.0 (40.2) | 134.2 (27.6) | 64.6 (16.2)
  Postoperative Day 3 (N=26,21,5) | 111.6 (43.9) | 123.5 (39.4) | 61.6 (20.8)
  Postoperative Day 4 (N=24,21,3) | 115.2 (63.0) | 123.5 (62.4) | 56.9 (29.3)
  Postoperative Day 5 (N=23,21,2) | 104.4 (47.4) | 108.6 (46.6) | 60.4 (41.9)
  Postoperative Day 6 (N=21,20,1) | 105.6 (44.0) | 106.6 (44.9) | 86.0 (0)
  Postoperative Day 7 (N=21,20,1) | 94.6 (46.7) | 96.1 (47.4) | 65.5 (0)
  Postoperative Day 8 (N=19,19,0) | 93.0 (45.8) | 93.0 (45.8) | 0 (0)
  Postoperative Day 9 (N=19,19,0) | 93.0 (46.9) | 93.0 (46.9) | 0 (0)
  Postoperative Day 10 (N=18,18,0) | 89.9 (49.7) | 89.9 (49.7) | 0 (0)
  Postoperative Day 11+ (N=15,15,0) | 75.3 (44.8) | 75.3 (44.8) | 0 (0)

10. Primary Outcome: Total Weight-Adjusted Dose of BAX326 Per Participant
Description: Assessed for the intra- and postoperative periods.
Time Frame: as for outcome 9
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: IU/kg
Units Other Than Participants: surgeries
Groups:
- Major Surgeries: Major surgery defined as surgeries which required moderate or deep sedation, general anesthesia, or major conduction blockade for patient comfort. It generally referred to major orthopedic (e.g., joint replacement), major abdominal, intracranial, cardiovascular, spinal and any other surgery which had a significant risk of large volume blood loss or blood loss into a confined anatomical space. Several tooth Minor surgeries.
Arm/Group | All Surgeries | Major Surgeries | Minor Surgeries
Number analyzed (Participants) | 28 | 17 | 13
Number analyzed (surgeries) | 38 | 21 | 17
IU/kg
  Intraoperative Period | 145 (70) | 191 (51) | 87 (43)
  Postoperative Period | 808 (766) | 1350 (617) | 138 (136)

11. Primary Outcome: Number of Units of Blood Product Transfused
Description: Blood product transfusions consisted of packed red blood cells (PRBC) or fresh frozen plasma (FFP) or both.
Time Frame: as for outcome 9
Population: Participants in the Full Analysis Set (exposed to BAX326 and provided suitable hemostatic efficacy data) who received blood product infusions during the intraoperative and/or postoperative period. Note: a unique participant could have more than one surgical procedure.
Measure: Mean (Standard Deviation); unit: units
Units Other Than Participants: surgery where blood transfusion given
Arm/Group | All Surgeries
Number analyzed (Participants) | 6
Number analyzed (surgery where blood transfusion given) | 6
units
  Intraoperative Period | 2.8 (1.2)
  Postoperative Period | 1.5 (0.7)

12. Primary Outcome: Volume of Blood Product Transfused
Description: Blood product transfusions consisted of packed red blood cells (PRBC) or fresh frozen plasma (FFP) or both.
Time Frame: as for outcome 9
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mL
Units Other Than Participants: surgery where blood transfusion given
Arm/Group | All Surgeries
Number analyzed (Participants) | 6
Number analyzed (surgery where blood transfusion given) | 6
mL
  Intraoperative period | 834.3 (358.7)
  Postoperative Period (2 surgeries) | 414.0 (227.7)

13. Primary Outcome: Safety: Number of Participants Who Developed Inhibitory Antibodies to Factor IX (FIX)
Time Frame: Throughout the study period (approximately 2 years 5 months)
Population: All participants in the Safety Analysis Set (participants exposed to BAX326 during the study). Note: a unique participant could be treated with BAX326 for more than one surgical procedure.
Measure: Number; unit: participants
Units Other Than Participants: treatments with BAX326 before surgery
Groups:
- Treatment With BAX326: All participants treated with BAX326 per planned surgical procedure and per unique participant. Data is reported as treatment with BAX326 per planned surgical procedure (including participants who discontinued in the study after treatment with BAX326 but before surgery was done) and per unique participants as a unique participant could be treated with BAX326 for more than one surgical procedure in this study.
Arm/Group | Treatment With BAX326
Number analyzed (Participants) | 30
Number analyzed (treatments with BAX326 before surgery) | 40
participants | 0

14. Primary Outcome: Safety: Number of Participants Who Developed Total Binding Antibodies to Factor IX (FIX)
Description: If there was more than 2-dilution increase as compared to pre-study level at screening.
Time Frame: Throughout the study period (approximately 2 years 5 months)
Population: as for outcome 13
Measure: Number; unit: participants
Units Other Than Participants: treatments with BAX326 before surgery
Arm/Group | Treatment With BAX326
Number analyzed (Participants) | 30
Number analyzed (treatments with BAX326 before surgery) | 40
participants | 0

15. Primary Outcome: Safety: Number of Adverse Events Related to BAX326
Time Frame: Throughout the study period (approximately 2 years 5 months)
Population: as for outcome 13
Measure: Number; unit: adverse events
Units Other Than Participants: treatments with BAX326 before surgery
Arm/Group | Treatment With BAX326
Number analyzed (Participants) | 30
Number analyzed (treatments with BAX326 before surgery) | 40
adverse events | 1

16. Primary Outcome: Safety: Occurence of a Thrombotic Event
Time Frame: Throughout the study period (approximately 2 years 5 months)
Population: as for outcome 13
Measure: Number; unit: surgeries
Units Other Than Participants: treatments with BAX326 before surgery
Arm/Group | Treatment With BAX326
Number analyzed (Participants) | 30
Number analyzed (treatments with BAX326 before surgery) | 40
surgeries | 0

17. Primary Outcome: Pre-Surgical Pharmacokinetics (PK): Area Under the Plasma Concentration Versus Time Curve (AUC) From 0 to 72 Hours Post-infusion Per Dose
Description: AUC0-72h (area under the plasma concentration/time curve from time 0 to 72 hours) was computed using the linear trapezoidal method. The concentration at 72 hours was interpolated from the two nearest sampling time points or extrapolated using the last quantifiable concentration and the terminal rate constant λz. λz was estimated from the slope of natural log-linear fitting to latter quantifiable concentrations, with largest adjusted R2.
Time Frame: Within 30 mins pre-infusion and post-infusion timepoints of 30 minutes, 6 hr, 24 hr, 48 hr and 72 hr
Population: Participants in the Full Analysis Set (exposed to BAX326 and provided data suitable for hemostatic efficacy analysis) who underwent a pre-surgical PK assessment in this study i.e.not participants who underwent a PK assessment in the pivotal study (250901). Note: a unique participant could have a pre-surgical PK assessment for more than one surgery.
Measure: Mean (Standard Deviation); unit: [IU•hour (hr)/dL] : IU/kg
Units Other Than Participants: pre-surgical PK assessments
Groups:
- Pre-surgical PK Assessment: A pre-surgical pharmacokinetic (PK) assessment was conducted for participants who had not undergone a PK assessment during the Pivotal study (Baxalta study 250901) before undergoing surgery in this study. Data is reported as pre-surgical PK assessment per surgical procedure as opposed to number of unique participants as a unique participant could have a pre-surgical PK assessment for more than one surgical procedure.
Arm/Group | Pre-surgical PK Assessment
Number analyzed (Participants) | 12
Number analyzed (pre-surgical PK assessments) | 12
[IU•hour (hr)/dL] : IU/kg | 18.48 (6.43)

18. Primary Outcome: Pre-Surgical Pharmacokinetics (PK): Total Area Under the Plasma Concentration Versus Time Curve Per Dose (Total AUC/Dose)
Description: Total AUC/Dose is also AUC0-inf (area under the plasma concentration/time curve from time 0 to infinity) and was defined as AUC0-t + Ct / λz, where t is the time of last quantifiable concentration, Ct is the last quantifiable concentration and λz is the terminal rate constant.
Time Frame: Within 30 mins pre-infusion and post-infusion timepoints of 30 minutes, 6 hr, 24 hr, 48 hr and 72 hr
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: [IU•hour (hr)/dL] : IU/kg
Units Other Than Participants: pre-surgical PK assessments
Arm/Group | Pre-surgical PK Assessment
Number analyzed (Participants) | 12
Number analyzed (pre-surgical PK assessments) | 12
[IU•hour (hr)/dL] : IU/kg | 20.60 (7.32)

19. Primary Outcome: Pre-Surgical Pharmacokinetics (PK): Mean Residence Time (MRT)
Description: The MRT is the average time that the study product stays in the body (or plasma) and is calculated as: AUMC 0-inf / AUC 0-inf, where AUMC 0-inf was determined in a similar manner as AUC 0-inf.
Time Frame: Within 30 mins pre-infusion and post-infusion timepoints of 30 minutes, 6 hr, 24 hr, 48 hr and 72 hr
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: hours (hr)
Units Other Than Participants: pre-surgical PK assessments
Arm/Group | Pre-surgical PK Assessment
Number analyzed (Participants) | 12
Number analyzed (pre-surgical PK assessments) | 12
hours (hr) | 27.17 (4.03)

20. Primary Outcome: Pre-Surgical Pharmacokinetics (PK): Factor IX (FIX) Clearance (CL)
Description: CL is the volume of plasma which is completely cleared of study product per unit time and is calculated as the dose divided by the total area under the curve from 0 to infinity (AUC0-inf).
Time Frame: Within 30 mins pre-infusion and post-infusion timepoints of 30 minutes, 6 hr, 24 hr, 48 hr and 72 hr
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: dL/(kg•hr)
Units Other Than Participants: pre-surgical PK assessments
Arm/Group | Pre-surgical PK Assessment
Number analyzed (Participants) | 12
Number analyzed (pre-surgical PK assessments) | 12
dL/(kg•hr) | 0.0523 (0.0126)

21. Primary Outcome: Pre-Surgical Pharmacokinetics (PK): Incremental Recovery (IR) at 30 Min
Description: IR was defined as (C post-infusion - C pre-infusion) / Dose, where C post-infusion is the measured concentration achieved at 30±5 minutes for pre-surgical PK.
Time Frame: Within 30 mins pre-infusion and post-infusion at 30 minutes
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: IU/dL : IU/kg
Units Other Than Participants: pre-surgical PK assessments
Arm/Group | Pre-surgical PK Assessment
Number analyzed (Participants) | 12
Number analyzed (pre-surgical PK assessments) | 12
IU/dL : IU/kg | 1.00 (0.29)

22. Primary Outcome: Pre-Surgical Pharmacokinetics (PK): Elimination Phase Half-life (T 1/2)
Description: T1/2 was determined as ln2 / λz.
Time Frame: Within 30 mins pre-infusion and post-infusion timepoints of 30 minutes, 6 hr, 24 hr, 48 hr and 72 hr
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: hours (hr)
Units Other Than Participants: pre-surgical PK assessments
Arm/Group | Pre-surgical PK Assessment
Number analyzed (Participants) | 12
Number analyzed (pre-surgical PK assessments) | 12
hours (hr) | 23.60 (3.60)

23. Primary Outcome: Pre-Surgical Pharmacokinetics (PK): Volume of Distribution at Steady State (Vss)
Description: Vss was computed as CL·MRT.
Time Frame: Within 30 mins pre-infusion and post-infusion timepoints of 30 minutes, 6 hr, 24 hr, 48 hr and 72 hr
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: dL/kg
Units Other Than Participants: pre-surgical PK assessments
Arm/Group | Pre-surgical PK Assessment
Number analyzed (Participants) | 12
Number analyzed (pre-surgical PK assessments) | 12
dL/kg | 1.41 (0.38)

24. Primary Outcome: Incremental Recovery (IR) at 15±5 Minutes Following Loading Dose Prior to Surgery
Description: IR was defined as (C post-infusion - C pre-infusion) / Dose, where C post-infusion is the measured concentration achieved at 15±5 minutes for the loading dose.
Time Frame: Within 60 minutes prior to surgery and 15 ± 5 minutes after loading dose/rebolus, if applicable.
Population: Participants in the Full Analysis Set (exposed to BAX326 and provided suitable hemostatic efficacy data) who provided data for incremental recovery (IR) after the loading dose prior to surgery. Note: a unique participant could have more than one surgical procedure.
Measure: Mean (Standard Deviation); unit: [IU/dL] : [IU/kg]
Units Other Than Participants: surgeries with IR data
Arm/Group | All Surgeries
Number analyzed (Participants) | 26
Number analyzed (surgeries with IR data) | 36
[IU/dL] : [IU/kg] | 0.910 (0.1787)

ADVERSE EVENTS:
Time Frame: Throughout the study period (approximately 2 years 5 months)
Groups:
- All Participants: All unique participants treated with BAX326 per planned surgical procedure.
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 10/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=30)
Post procedural swelling (Injury, poisoning and procedural complications) | 3
Procedural pain (Injury, poisoning and procedural complications) | 7
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 3
Thrombocytosis (Blood and lymphatic system disorders) | 4

LIMITATIONS AND CAVEATS:
Data provided for surgical procedures, treatments with BAX326 etc. and for unique participants (one unique participant could undergo more than one surgical procedure).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Baxalta's agreements with PIs may vary per requirements of individual PI, but contain common elements. For this study, results may not be published without prior written approval of the Sponsor.